CLINICAL TRIAL: NCT06837194
Title: The Efficacy of WMT Combined with Nutritional Support in the Treatment of Malnutrition Complicated by Gastroptosis: a Real-World Study
Brief Title: Washed Microbiota Transplantation Combined with Enteral Nutrition for Gastroptosis
Status: Recruiting | Type: Observational
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Other Study IDs: WMT-gastroptosis
Record Dates: First submitted 2025-02-10; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Gastroptosis; Malnutrition
Keywords: washed microbiota transplantation; microbiota medicine; Gastroptosis; malnutrition; enteral nutrition; Transendoscopic Enteral Tubing
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Years
Biospecimen Retention: Samples Without DNA — Feces, urine and blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observation Group: Washed microbiota transplantation refers to the infusion of washed microbiota from healthy donor into patients' gastrointestinal tract. Participants will receive three doses of WMT and enteral nutrition for three months for gastroptosis.

SUMMARY:
This is a observational study to explore the efficacy and safety of washed microbiota transplantation (WMT) combined with nutritional support for gastroptosis patients

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to enter the study:

  1. Clinically diagnosed with gastroptosis;
  2. Meets the diagnostic criteria for malnutrition (fulfilling any one of the following two criteria):

     * Weight loss (weight loss >5% within the last 6 months or >10% over more than 6 months);

       * Low BMI (BMI <18.5 kg/m² for individuals <70 years old; BMI <20 kg/m² for individuals ≥70 years old);
  3. Males aged ≥18 years and non-pregnant, non-lactating females aged ≥18 years;
  4. Willing to voluntarily sign a written informed consent form and agrees to follow medical advice for regular follow-up examinations and monitoring after the completion of treatment.

Exclusion Criteria:

* Subjects meeting any of the following exclusion criteria must be excluded from the study:

  1. Patients with severe depression, anxiety, or cognitive impairment that affects normal physician-patient communication and treatment planning;
  2. Patients with poor compliance who cannot accept treatment regimens such as nasogastric enteral nutrition;
  3. Anticipated survival time <3 months;
  4. Clinically significant cardiovascular diseases, including heart failure (NYHA Class III-IV), uncontrolled coronary artery disease, cardiomyopathy, arrhythmia, history of myocardial infarction, hemodynamic instability at enrollment, unstable vital signs, or anticipated risk events during treatment;
  5. Poor pulmonary function deemed by investigators to impact study treatment (e.g., acute exacerbation of COPD or requirement for long-term oral/intravenous corticosteroids [excluding inhaled corticosteroids]);
  6. Active severe clinical infections (> Grade 2 per NCI-CTCAE v5.0), including patients with intestinal fungal, viral, or tuberculosis infections;
  7. Inability to cooperate with intestinal tube placement or contraindications to intestinal tube placement;
  8. Use of medications affecting or modulating gut microbiota within the past 48 hours;
  9. Lack of legal capacity or restricted legal capacity;
  10. Hematologic disorders unsuitable for blood draw examinations;
  11. Other severe medical conditions deemed by investigators to preclude patient enrollment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years old with malnutrition and gastroptosis
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of gastroptosis with degree relief after the procedure. | baseline, 12 weeks post transplantation
  Detailed evaluation content of efficacy rate of degree: The ultrasound examination was divided into three levels of light, medium and heavy according to the specific value of the middle gastric angle below Iliac spines are connected, defined as a reduction of at least 50% in value or a reduction of degree.

SECONDARY OUTCOMES:
change of the third lumbar vertebrae skeletal muscle mass and height | baseline, 12 weeks post transplantation
  The third lumbar vertebrae skeletal muscle mass represents the sum of the cross-sectional areas of the skeletal muscles at the L3 level, including the psoas major, the erector spinae, the quadratus lumborum, the musculus transversus abdominis, the obliquus externus abdominis and the obliquus internus abdominis. Skeletal muscle mass and height will be combined to report the third lumbar vertebrae skeletal muscle mass index(L3 SMI) in cm^2/m^2.
change of weight and height | baseline, 4 weeks, 8 weeks, 12 weeks post transplantation
  Weight and height will be combined to report BMI in kg/m^2.
change of the Gastrointestinal Symptom Rating Scale(GSRS) | baseline, 4 weeks, 8 weeks, 12 weeks post transplantation
  GSRS is a 13-item test to make a comprehensive assessment of common gastrointestinal symptom and each item receives a value from 0 to 3, with higher value indicating worse gastrointestinal condition.
The extent of change observed in Gastroparesis Cardinal Symptom Index(GCSI)of participants | baseline, 4 weeks, 8 weeks, 12 weeks post transplantation
  The GCSI consists of nine items and three subscales to measure symptoms related to gastroparesis. The nausea/vomiting subscale consists of the following three items: nausea, retching, and vomiting. The postprandial fullness/early satiety subscale consists of the following four items: stomach fullness, inability to finish a normal-sized meal, feeling excessively full after meals, and loss of appetite.
The results of gastric fitted emptying rate data for 2 hours or 4 hours in the gastric emptying experiment with nuclide imaging | baseline, 12 weeks post transplantation
change of the 5-level EuroQoL Group's 5-dimension (EQ-5D-5L) | baseline, 4 weeks, 8 weeks, 12 weeks post transplantation
  EQ-5D-5L is a 5-dimension questionnaire measuring health state and each dimension represents the level from 1 to 5, with higher level indicating worse health state.
change of the Pittsburgh Sleep Quality Index (PSQI) | baseline, 4 weeks, 8 weeks, 12 weeks post transplantation
  PSQI is a self-rated questionnaire which assesses sleep quality over a 1-month time interval. Nineteen items generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for seven components yields one global score, with higher score indicating worse sleep quality.
change of the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) | baseline, 4 weeks, 8 weeks, 12 weeks post transplantation
  FACIT-Fatigue is a 13-item test measuring fatigue and each item receives a value from 0 to 4, with higher value indicating worse fatigue state.
The extent of change observed in gastrointestinal ultrasound (GIUS) of participants | baseline, 12 weeks post transplantation
  The half gastric emptying time will be evaluated by GIUS.
The extent of change observed in transcranial Doppler (TCD) of participants | baseline, 12 weeks post transplantation
  TCD was used to evaluate the degree of continuity of echo in the nucleus suture in patients, and echoic discontinuity represented the possibility of anxiety and depression.
change of the Hamilton Anxiety Scale(HAMA) | baseline, 4 weeks, 8 weeks, 12 weeks post transplantation
  Hamilton Anxiety Scale is a 14-item test measuring anxiety and each item receives a value from 0 to 4, with higher value indicating worse anxiety state.
change of the Hamilton Depression Scale(HAMD） | baseline, 4 weeks, 8 weeks, 12 weeks post transplantation
  Hamilton Depression Scale is a 17-item test measuring depression and each item receives a value from 0 to 4, with higher value indicating worse depression state.
change of insulin-like growth factor I(IGF-I) | baseline, 12 weeks post transplantation
  Blood is tested for Insulin-like growth factor I.
change of albumin and Prealbumin | baseline, 12 weeks post transplantation
  Blood is tested for albumin and Prealbumin.
change of cytokine | baseline, 12 weeks post transplantation
  Blood is tested for IL-1β、IL-2、IL-4、IL-5、IL-6、IL-8、IL-10、IL-12p70、IL-17、TNF-α、IFN-γ、IFN-α.
The changes in gut microbiota composition and metabolites before and after treatment | baseline, 12 weeks post transplantation
  The 16s-RNA or meta-analysis of gut microbiota will be used.
the incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0 | 12 weeks post transplantation
  The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Department of Microbiota Medicine & Medical Centre for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang F, Cui B, He X, Nie Y, Wu K, Fan D; FMT-standardization Study Group. Microbiota transplantation: concept, methodology and strategy for its modernization. Protein Cell. 2018 May;9(5):462-473. doi: 10.1007/s13238-018-0541-8. Epub 2018 Apr 24. PMID 29691757
- [Background] Peng Z, Xiang J, He Z, Zhang T, Xu L, Cui B, Li P, Huang G, Ji G, Nie Y, Wu K, Fan D, Zhang F. Colonic transendoscopic enteral tubing: A novel way of transplanting fecal microbiota. Endosc Int Open. 2016 Jun;4(6):E610-3. doi: 10.1055/s-0042-105205. Epub 2016 Apr 28. PMID 27556065
- [Background] Quince C, Ijaz UZ, Loman N, Eren AM, Saulnier D, Russell J, Haig SJ, Calus ST, Quick J, Barclay A, Bertz M, Blaut M, Hansen R, McGrogan P, Russell RK, Edwards CA, Gerasimidis K. Extensive Modulation of the Fecal Metagenome in Children With Crohn's Disease During Exclusive Enteral Nutrition. Am J Gastroenterol. 2015 Dec;110(12):1718-29; quiz 1730. doi: 10.1038/ajg.2015.357. Epub 2015 Nov 3. PMID 26526081
- [Background] Xiang L, Yu Y, Ding X, Zhang H, Wen Q, Cui B, Zhang F. Exclusive Enteral Nutrition Plus Immediate vs. Delayed Washed Microbiota Transplantation in Crohn's Disease With Malnutrition: A Randomized Pilot Study. Front Med (Lausanne). 2021 Oct 22;8:666062. doi: 10.3389/fmed.2021.666062. eCollection 2021. PMID 34746161
- [Background] Fernandes ND, Murphy SA. Gastroptosis: An Uncommon Cause for a Deep Nasogastric Tube. Clin Gastroenterol Hepatol. 2021 Jun;19(6):A23. doi: 10.1016/j.cgh.2020.04.016. Epub 2020 Apr 11. No abstract available. PMID 32289543
- [Background] Xu LC, Garcia JC. Gastroptosis in a young woman. Gastrointest Endosc. 2024 Mar;99(3):454-455. doi: 10.1016/j.gie.2023.10.006. Epub 2023 Oct 5. No abstract available. PMID 37804872